CLINICAL TRIAL: NCT00661479
Title: An Exploratory Study to Evaluate the Safety of Brimonidine Intravitreal Implant in Patients With Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 190342-028D
Record Dates: First submitted 2007-10-29; First posted 2008-04-18 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-03

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Brimonidine Tartrate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 400 µg Brimonidine Tartrate Implant Group B (Experimental): 400 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1.
  Interventions: Drug: 400 µg Brimonidine Tartrate Implant; Other: Sham (no implant)
- 200 µg Brimonidine Tartrate Implant Group B (Experimental): 200 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1.
  Interventions: Drug: 200 µg Brimonidine Tartrate Implant; Other: Sham (no implant)
- 100 µg Brimonidine Tartrate Implant Group B (Experimental): 100 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1.
  Interventions: Drug: 100 µg Brimonidine Tartrate Implant; Other: Sham (no implant)
- 100 µg Brimonidine Tartrate Implant Group A (Experimental): 100 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1.
  Interventions: Drug: 100 µg Brimonidine Tartrate Implant; Other: Sham (no implant)

INTERVENTIONS:
Drug: 400 µg Brimonidine Tartrate Implant — 400 µg brimonidine tartrate implant in the study eye on Day 1.
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 400 µg Brimonidine Tartrate Implant Group B
Drug: 200 µg Brimonidine Tartrate Implant — 200 µg brimonidine tartrate implant in the study eye on Day 1.
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 200 µg Brimonidine Tartrate Implant Group B
Drug: 100 µg Brimonidine Tartrate Implant — 100 µg brimonidine tartrate implant in the study eye on Day 1.
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 100 µg Brimonidine Tartrate Implant Group A; 100 µg Brimonidine Tartrate Implant Group B
Other: Sham (no implant) — Sham in the fellow eye on Day 1.

SUMMARY:
This exploratory, 12-month, ascending-dose study will evaluate the safety and effects on visual function of a single injection of Brimonidine intravitreal implant in one eye of patients with Retinitis Pigmentosa.

ELIGIBILITY:
Inclusion Criteria:

* Retinitis Pigmentosa in both eyes
* Visual acuity between 20/40 to count fingers

Exclusion Criteria:

* Growth of new blood vessels in the eye
* Any intraocular surgery or laser in either eye in the last 6 months prior to Screening visit or between the Screening visit and Day 1
* Any ocular disease that can interfere with diagnosis and or assessment of disease progression
* Significant near-sightedness
* HIV
* Female patients who are pregnant, nursing, or planning pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Arlington, Texas, United States
- Paris, France
- Tübingen, Germany
- Coimbra, Portugal

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were stratified by Best Corrected Visual Acuity (BCVA). Patients assigned to Group A had a BCVA of 20/320. Patients assigned to Group B had a BCVA worse than 20/40 and better than 20/320. Patients in Group A were randomized and treated prior to initiating enrollment in Group B. No patients from Group A participated in Group B.
Period: Overall Study
Arm/Group | 400 µg Brimonidine Tartrate Implant Group B | 200 µg Brimonidine Tartrate Implant Group B | 100 µg Brimonidine Tartrate Implant Group B | 100 µg Brimonidine Tartrate Implant Group A
Started | 12 | 3 | 3 | 3
Completed | 12 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 µg Brimonidine Tartrate Implant Group B | 200 µg Brimonidine Tartrate Implant Group B | 100 µg Brimonidine Tartrate Implant Group B | 100 µg Brimonidine Tartrate Implant Group A | Total
Number analyzed (Participants) | 12 | 3 | 3 | 3 | 21
Age Continuous [Mean (Standard Deviation); unit: Years] | 46.3 (18.70) | 56.3 (6.03) | 48.7 (4.04) | 69.0 (5.29) | 51.3 (16.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 0 | 9
  Male | 7 | 2 | 0 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening.
Time Frame: Baseline, Month 6
Population: Safety Population: all patients treated on Day 1
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | 400 µg Brimonidine Tartrate Implant Group B | 200 µg Brimonidine Tartrate Implant Group B | 100 µg Brimonidine Tartrate Implant Group B | 100 µg Brimonidine Tartrate Implant Group A
Number analyzed (Participants) | 12 | 3 | 3 | 3
Number of Letters Read Correctly
  Baseline | 48.5 (14.61) | 51.0 (14.18) | 52.7 (3.79) | 4.0 (3.46)
  Change from Baseline at Month 6 | 3.2 (4.41) | -1.3 (4.04) | 3.3 (8.50) | 0.3 (3.79)

2. Secondary Outcome: Change From Baseline in Contrast Sensitivity in the Study Eye
Description: Change from baseline in contrast sensitivity in the study eye is measured using a Pelli-Robson contrast sensitivity chart at 1 meter. The contrast sensitivity chart contains letters that are darkest at the top and then get progressively lighter. Scores range from 0 to 48 and are based on the number of letters read correctly. A negative change from baseline indicates a worsening in contrast sensitivity and a positive change from baseline indicates an improvement.
Time Frame: Baseline, Month 6
Population: Safety Population: all patients treated on Day 1
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | 400 µg Brimonidine Tartrate Implant Group B | 200 µg Brimonidine Tartrate Implant Group B | 100 µg Brimonidine Tartrate Implant Group B | 100 µg Brimonidine Tartrate Implant Group A
Number analyzed (Participants) | 12 | 3 | 3 | 3
Number of Letters Read Correctly
  Baseline | 15.5 (8.48) | 18.0 (7.21) | 22.3 (1.53) | 3.0 (3.46)
  Change from Baseline at Month 6 | 0.8 (4.86) | -0.3 (5.86) | 4.3 (1.15) | -2.0 (1.73)

ADVERSE EVENTS:
Description: For Ocular AEs, only those occurring in the study eye are reported in the "Other Adverse Events" section. For SAEs, all ocular events were reported, regardless of eye.
Groups:
- 100 µg Brimonidine Tartrate Implant Groups A and B: 100 µg brimonidine tartrate implant in the study eye and sham in the fellow eye on Day 1.
Arm/Group | 400 µg Brimonidine Tartrate Implant Group B | 200 µg Brimonidine Tartrate Implant Group B | 100 µg Brimonidine Tartrate Implant Groups A and B
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 11/12 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 µg Brimonidine Tartrate Implant Group B (N=12) | 200 µg Brimonidine Tartrate Implant Group B (N=3) | 100 µg Brimonidine Tartrate Implant Groups A and B (N=6)
Syncope (Nervous system disorders) | 1 | 0 | 0
Myelitis (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 400 µg Brimonidine Tartrate Implant Group B (N=12) | 200 µg Brimonidine Tartrate Implant Group B (N=3) | 100 µg Brimonidine Tartrate Implant Groups A and B (N=6)
Conjunctival Haemorrhage (Eye disorders) | 5 | 2 | 1
Conjunctival Hyperaemia (Eye disorders) | 5 | 3 | 5
Foreign Body Sensation in Eyes (Eye disorders) | 3 | 0 | 1
Ocular Discomfort (Eye disorders) | 3 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 2
Fatigue (General disorders) | 2 | 0 | 0
Glare (Eye disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Eye Pain (Eye disorders) | 2 | 0 | 2
Conjunctival Oedema (Eye disorders) | 2 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Colour Blindness (Congenital, familial and genetic disorders) | 1 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dry Eye (Eye disorders) | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1/7 | 0/2 | 0/3
Eye Irritation (Eye disorders) | 1 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Lacrimation Increased (Eye disorders) | 1 | 0 | 0
Ligament Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Visual Disturbance (Eye disorders) | 1 | 0 | 0
Abnormal Sensation in Eye (Eye disorders) | 0 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myelitis (Nervous system disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Prostate Infection (Infections and infestations) | 0/7 | 0/2 | 1/3
Renal Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Restless Legs Syndrome (Nervous system disorders) | 0 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1
Vitreous Floaters (Eye disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.